CLINICAL TRIAL: NCT02761408
Title: Correlation Between Radiation Dermatitis/Mucositis and ALDH2 Mutation in Taiwanese Head and Neck Cancer
Brief Title: ALDH2 Mutation in Taiwanese Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-03-008AC
Record Dates: First submitted 2016-04-26; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Dermatitis; Mucositis
Keywords: Head and neck cancer; Asian; ALDH2
MeSH Terms: conditions — Dermatitis; Mucositis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effect of ALDH2 mutation in radiation associating dermatitis or mucositis in head and neck cancer patients who accept chemoradiation therapy

DETAILED DESCRIPTION:
* One-site audit. The enrolled subject is confirmed by PIs

  ◦◦Source data is compared to external data sources medical records, either paper or electronic case report forms.
* NCI CTCAE v5.0 for AE records
* Patient recruitment according to inclusion criteria: 1. Newly diagnosed locally head and neck squamous cell carcinoma; 2. Apply for primary chemoradiation or adjuvant chemoradiation; 3. Signed informed consent
* Sample size assessment: 60 subjects will be included in one year for total 120 subjects
* Missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results
* Fisher's exact test is for category comparison. Kaplan-Meier analysis is for survival analysis. AE grades will be analyzed according to NCI guideline. Two-side p < 0.05 is suggested significant.

ELIGIBILITY:
Inclusion Criteria:

* Age >20, <70
* Newly diagnosed head and neck squamous cell carcinoma
* Tissue proved
* Signed informed consent
* Suitable for chemoradiation

Exclusion Criteria:

* Uncontrolled underlying diseases
* Allergy to chemotherapy
* Uncontrolled skin diseases or mucosa diseases
* Previously radiation therapy over head and neck
* Combined with other cancer currently

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced Taiwanese head and neck squamous cell carcinoma patients who intend to accept primary chemoradiation or surgery with adjuvant chemoradiation, without previous treatment
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAEv5.0 | 6 months after the end of the study
  The side effects of each participant will be recorded accoiding to CTCAEv5.0 during the whole course of chemoradiation, by indicated physicians regularly

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Wei Wang, MD, Principal Investigator — Cancer Center, Taipei Veterans General Hospital
Locations (1):
- Cancer Center, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No